CLINICAL TRIAL: NCT06489964
Title: Addressing the Problem of Recommended But Unfunded Vaccines Through a Co-payment Mechanism in Pharmacies
Brief Title: Addressing Unfunded Vaccines Through a Co-payment Mechanism in Pharmacies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Immunization Research Network (Network)
Collaborators: Dalhousie University (Other); AstraZeneca (Industry); GlaxoSmithKline (Industry); Canadian Center for Vaccinology (Other)
Responsible Party: Principal Investigator, Emily Black, Associate Professor, Canadian Immunization Research Network
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SH37
Record Dates: First submitted 2024-05-30; First posted 2024-07-08 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Preventable Disease, Vaccine
MeSH Terms: conditions — Vaccine-Preventable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Community Pharmacy Sites (Step 1) (Other): A pharmacy site in Nova Scotia and Ontario will be randomly assigned to pilot Step 1 of the co-payment model for the duration of the pilot study.
  Interventions: Other: Co-payment Model - Step 1
- Community Pharmacy Sites (Step 2) (Other): A pharmacy site in Nova Scotia and Ontario will be randomly assigned to pilot Step 2 of the co-payment model for the duration of the pilot study.
  Interventions: Other: Co-payment Model - Step 2
- Community Pharmacy Sites (Step 3) (Other): A pharmacy site in Nova Scotia and Ontario will be randomly assigned to pilot Step 3 of the co-payment model for the duration of the pilot study.
  Interventions: Other: Co-payment Model - Step 3
- Community Pharmacy Sites (Step 4) (Other): A pharmacy site in Nova Scotia and Ontario will be randomly assigned to pilot Step 4 of the co-payment model for the duration of the pilot study.
  Interventions: Other: Co-payment Model - Step 4

INTERVENTIONS:
Other: Co-payment Model - Step 1 — Step 1 of the co-payment model: A pharmacy site from Nova Scotia and Ontario will be randomly assigned to this step where the study will cover the administration service fee (approximately $35.00) and the participant will pay 100% of the vaccine cost out-of-pocket for the eligible vaccine. The vaccines will include FluMist Quadrivalent, Shingrix, and Abrysvo or Arexvy.
  Arms: Community Pharmacy Sites (Step 1)
Other: Co-payment Model - Step 2 — Step 2 of the co-payment model: A pharmacy site from Nova Scotia and Ontario will be randomly assigned to this step where the study will cover 50% of the vaccine cost plus the administration service fee and the participant will pay 50% of the vaccine cost out-of-pocket. The vaccines will include FluMist Quadrivalent, Shingrix, Abrysvo or Arexvy.
  Arms: Community Pharmacy Sites (Step 2)
Other: Co-payment Model - Step 3 — Step 3 of the co-payment model: A pharmacy site from Nova Scotia and Ontario will be randomly assigned to this step where the study will cover 75% of the vaccine cost plus the administration service fee and the participant will pay 25% of the vaccine cost out-of-pocket. The vaccines will include FluMist Quadrivalent, Shingrix, and Abrysvo or Arexvy.
  Arms: Community Pharmacy Sites (Step 3)
Other: Co-payment Model - Step 4 — Step 4 of the co-payment model: A pharmacy site from Nova Scotia and Ontario will be randomly assigned to this step where the study will cover 100% of the vaccine cost plus the administration service fee and the participant will pay 0% of the vaccine cost. The vaccines will include FluMist Quadrivalent, Shingrix, and Abrysvo or Arexvy.
  Arms: Community Pharmacy Sites (Step 4)

SUMMARY:
The goal of this pilot demonstration and evaluation project is to determine the acceptability and feasibility of a co-payment model among the public and providers and assess whether a co-payment model in community pharmacies in Nova Scotia and Ontario increases the accessibility and uptake of recommended but unfunded vaccines. The research questions that guided the development of this study are:

* What is the feasibility of implementing a co-payment model for recommended but unfunded vaccines in community pharmacies?
* To what extent is a co-payment model for recommended but unfunded vaccines perceived as acceptable to community pharmacists and the public?

A co-payment model will be piloted at a maximum of 8 select community pharmacy sites in Nova Scotia (n=4 sites) and Ontario (n=4 sites). Each community pharmacy site will be randomly assigned to pilot one of the steps of the co-payment model for the duration of the demonstration project. At the end of the pilot study, participating pharmacy providers will be asked to complete an online survey about their experiences in implementing the co-payment model into their pharmacy. As part of the co-payment model, recruited members of the public (participants) will choose to receive the vaccine (if eligible) at a reduced cost either for themselves or their dependent (e.g., incapable minor or adult), as part of routine care (following standard pharmacy practice). After receiving the vaccine, the participant will complete an online survey exploring their thoughts on the co-payment model, their satisfaction with the co-payment model, their perception on vaccines in general, and their demographics (such as gender, age, education, race/ethnicity).

DETAILED DESCRIPTION:
While the National Advisory Committee on Immunization (NACI) provides vaccine recommendations, it is the responsibility of provinces and territories in Canada to decide which vaccine programs they will support and implement publicly. Some vaccines recommended by NACI are not publicly funded in Canada and require out-of-pocket pay or private health insurance plans. This lack of public funding may be a factor contributing to low vaccine uptake. Cost-related barriers are also important concerns among prescribers who tend to be hesitant in recommending vaccines that are not publicly funded due to issues with patient affordability. Pharmacy professionals (in some jurisdictions) across Canada are increasingly taking a dominant role in administering certain publicly funded vaccines such as influenza and COVID-19. However, administration of other recommended and publicly funded immunizations have been limited in many jurisdictions, and pharmacy services providing unfunded vaccines are underutilized.

Current publicly funded immunization programs have proven to be cost-effective for the health care system; however, assessing the economic impact of vaccines takes time, resulting in recommended vaccines not being funded for some or all individuals. This economic impact of the initial, upfront costs of introducing a vaccine program can be financially prohibitive, acting as a major barrier to having vaccinations covered through public funding. As a result, introducing a co-payment system for recommended but unfunded vaccines may help mitigate the perception that these vaccines are of lesser importance, especially if the government is covering a portion of the vaccine and administration fees. A flexible co-payment model, where the costs are shared between the patient or their private insurance and the government, until full funding becomes available, could potentially offer a solution to enhance immunization rates for these vaccines.

In this Pilot Demonstration and Evaluation Project, the investigators propose to better understand potential solutions to cost-related barriers that limit uptake of recommended but unfunded vaccines, with alternative funding models being one possible solution. Implementation of a co-payment funding model within community pharmacies will be piloted at select community pharmacies in Nova Scotia and Ontario where pharmacy providers will prescribe and administer recommended but unfunded vaccines, as part of routine care. Electronic surveys will assess public and provider satisfaction with the model and the number of people vaccinated before and during the pilot demonstration will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Community Pharmacy Sites: Inclusion criteria for the selection of the community pharmacies will include volume of prescriptions (e.g., how busy the site it), stable pharmacy patients (e.g., patients who consistently use the same pharmacy), availability and interest of community pharmacies and community pharmacy professionals, sufficient numbers of pharmacy professionals qualified to provide vaccinations, and lack of substantial health care spill over to adjacent communities. Spill over is defined as a pattern of health-care utilization where the public regularly receive care at different regional health centres. Communities will be geographically separated to minimize potential spill over. Based on this inclusion criteria, one pharmacy from the four health zones in Nova Scotia will be selected to implement the co-payment model within their community pharmacy, while a mix of urban and rural pharmacies in Ontario will be selected to implement the co-payment model.
* Members of the Public: The participating pilot pharmacies will recruit through targeted screening members of the public who meet the vaccine-specific eligibility criteria or their substitute decision-makers for those who lack capacity to consent. Any members of the public or the substitute decision-maker who consents to participate will be eligible until the maximum number of participants we aim to recruit has been achieved. Eligible members of the public will receive the vaccines based on NACI recommendations for each product as part of routine care.
* Recommended but Unfunded Vaccines: FluMist Quadrivalent: An age-appropriate quadrivalent influenza should be used in children (2 to 17 years) without contraindications or precautions; Shingrix Vaccine: Adults 50 to 64 years of age in Nova Scotia or 50 years of age or older in Ontario without contraindications or adults 18 years of age or older if immunocompromised; and Abrysvo or Arexvy (RSV) vaccine: Adults 50 years of age or older (Arexvy) or 60 years of age and older (Abrysvo) who are at increased risk of severe RSV disease. Note: The eligibility criteria for each vaccine product may be revised during the pilot study if there are any changes in vaccine recommendations and/or funding status in Nova Scotia or Ontario.

Exclusion Criteria:

* FluMist Quadrivalent: should not be used in children or adolescents for whom it is contraindicated or for whom there are warnings and precautions; should not be used in children or adolescents already adequately immunized against influenza; not recommended for pregnant individuals, health care workers, and adult 18 to 59 years old with specific chronic health conditions; adults 60 to 64 and 65 years and old, as this vaccine is not authorized for use in these age groups; pediatric children (2 to 17 years) of the participating pharmacies who already have private insurance coverage to cover all (or most) of the FluMist vaccine will be excluded from taking part in this study.
* Shingrix: Persons with active herpes zoster (HZ) should not be immunized with HZ vaccine; should not be used in individuals already adequately immunized against HZ; adults 65 years of age or older in Nova Scotia, as this vaccine is publicly funded for this age group; adults 65 to 70 years of age in Ontario, as this vaccine is publicly funded for this age group; and adults (50 to 64 years old in Nova Scotia and 50 years of age or older in Ontario) of the participating pharmacies who already have private insurance coverage to cover all (or most) of the Shingrix vaccine will be excluded from taking part in this study.
* Abrysvo or Arexvy (RSV): Persons under the age 50 years should not be immunized with RSV vaccine (exception is use of Abrysvo in pregnancy), as it is not authorized for use in this age group; should not be used in individuals already adequately immunized against RSV; adults 60 years and older in Nova Scotia living in long-term care facilities or in hospital awaiting long-term care placement, as this vaccine is publicly funded for this age group; high-risk older adults (aged 60 years and older) in Ontario (e.g., residents of long-term care homes, Elder Care Lodges, or retirement homes; patients in hospital receiving alternate level of care; patients receiving hemodialysis or peritoneal dialysis; recipients of solid organ or hematopoietic stem cell transplants; individuals experiencing homelessness; and individuals who identify as First Nations, Inuit, or Métis); and adults (≥ 50 years of age (AREXVY) or 60 years of age (Abrysvo) at increased risk of severe RSV disease) of the participating pharmacies who already have private insurance coverage to cover all (or most) of the RSV vaccine will be excluded from taking part in this study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Evaluating Acceptability of Implementing of a Co-Payment Model within Community Pharmacies through Surveys with Members of the Public and Community Pharmacy Providers | 6 months
  After choosing to receive a vaccine at a reduced cost either for themselves or their dependent (e.g., incapable minor or adult) as part of the co-payment model, participants will be asked to complete an online survey about their participation in the co-payment model. At the end of the pilot study, pharmacy providers who take part in the study will be asked to complete an online survey about implementing the co-payment model within their pharmacy practice. The surveys have been developed based on the Theoretical Framework of Acceptability and include questions on the acceptability of the co-payment model. To evaluate acceptability of implementing a co-payment model within community pharmacies, data from the public and provider surveys will be analyzed using basic descriptive statistics. Factors that may influence acceptability of the co-payment model (e.g. geography, gender, age, socioeconomic status, ethnicity, and cost) will also be assessed.
Evaluating Feasibility of Implementing a Co-Payment Model within Community Pharmacies through Surveys with Members of the Public and Community Pharmacy Providers | 6 months
  After choosing to receive a vaccine at a reduced cost either for themselves or their dependent (e.g., incapable minor or adult) as part of the co-payment model, participants will be asked to complete an online survey about their participation in the co-payment model. At the end of the pilot study, pharmacy providers who take part in the study will be asked to complete an online survey about implementing the co-payment model within their pharmacy practice. The surveys have been developed based on the Theoretical Framework of Acceptability and include questions on the feasibility of the co-payment model. To evaluate the feasibility of implementing a co-payment model within community pharmacies, data from the public and provider surveys will be analyzed using basic descriptive statistics. Factors that may influence feasibility of the co-payment model such as geography (urban vs. rural), gender, age, socioeconomic status, ethnicity, and cost to the patient will also be assessed.

SECONDARY OUTCOMES:
Descriptively report on the number of vaccines administered at participating community pharmacy sites before and during implementation of the co-payment model | 30 months
  To compare the number of people vaccinated before and during the pilot demonstration will be measured using pharmacy-generated reports of the number of vaccines administered at participating community pharmacies before and during implementation of the co-payment model.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Black, PharmD, Principal Investigator — Dalhousie University
Locations (2):
- Canada (2):
  - Dalhousie University, Halifax, Nova Scotia
  - University of Waterloo, Kitchener, Ontario

IPD SHARING:
Plan to Share IPD: No